CLINICAL TRIAL: NCT00761956
Title: Prospective Randomized Multicenter Study of NexGen CR-Flex Knee
Brief Title: A Study to Compare the NexGen CR and CR-Flex Knee Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04-300
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2012-07-16 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-06

CONDITIONS: Total Knee Arthroplasty; Osteoarthritis
Keywords: Total Knee Arthroplasty; Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Study arm will consist of patients that are treated with the NexGen CR-Flex Fixed Bearing Knee.
  Interventions: Device: NexGen CR-Flex Fixed Bearing Knee
- 2 (Active Comparator): Study arm will consist of patients that are treated with the NexGen CR Knee.
  Interventions: Device: NexGen CR Knee

INTERVENTIONS:
Device: NexGen CR-Flex Fixed Bearing Knee — NexGen CR-Flex Fixed Bearing femoral component
  Other Names: CR-Flex Knee
  Arms: 1
Device: NexGen CR Knee — NexGen Complete Knee Solution Cruciate Retaining femoral component
  Other Names: CR Knee
  Arms: 2

SUMMARY:
The purpose of this study is to test for significant differences in functional outcomes, specifically pre-operative ROM and post-operative ROM obtained by using a NexGen CR versus a NexGen CR-Flex knee implant. Specifically, it is predicted that an increase in post-operative range of motion will be experienced by patients treated with the NexGen CR-Flex knee implant.

DETAILED DESCRIPTION:
This study will compare the clinical results of the NexGen CR femoral component with the higher flexion potential of the NexGen CR-Flex femoral component in all patients with degenerative joint disease that require total knee arthroplasty. The primary variable of interest is post-operative range of motion achieved with the two devices, which are implanted with slightly different surgical techniques in patients who may also be subjected to different rehabilitation programs depending on the device they are assigned.

ELIGIBILITY:
Inclusion Criteria:

* Age, 21-80 years
* Sex, Male and Females will be included
* BMI less than or equal to 39
* Stable Health, the patient would be able to undergo surgery and participate in a follow-up program based on physical examination and medical history.
* Patient is willing and able to cooperate in follow-up therapy.
* Patient exhibits pre-operative radiographic evidenced of joint degeneration consistent with TKA that cannot be treated in non-operative fashion.
* Patient has stable and functional posterior cruciate and collateral ligaments.
* Patient has potential to perform higher than average range of motion activities.
* Operative side range of motion flexion greater than or equal to 120 degrees.
* Severe knee pain and disability due to degenerative joint disease.
* Patient or patient's legal representative has signed the Informed Consent form.

Exclusion Criteria:

* Previous history of infection in the affected joint.
* Previously failed knee endoprosthesis of any kind.
* Charcot joint disease or other severe neurosensory deficits.
* Previous patellectomy
* Patient is skeletally immature.
* Grossly insufficient femoral or tibial bone stock.
* Patient is pregnant.
* Varus or valgus deformity greater than 20 degrees.
* Fixed flexion deformity greater than 15 degrees.
* Previous high tibial osteotomy.
* Previous femoral osteotomy.
* Patient is a poor compliance risk, currently treated for ethanol or drug abuse, physical or mental handicap, etc.
* Loss of musculature or absence of musculoligamentous supporting structures required for adequate soft tissue balance.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2004-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Dickinson Medical Group, LLC, Milford, Delaware
  - University of Chicago Hospital, Chicago, Illinois
  - Rockford Orthopedic Associates, Rockford, Illinois
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Orthopaedic Associates of Grand Rapids, PC, Grand Rapids, Michigan
  - Pinehurst Surgical Center, Pinehurst, North Carolina
  - Slocum Orthopedics, PC, Eugene, Oregon
  - The Orthopedic Group, Clairton, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between 2004 and 2008 at a total of 15 sites throughout the USA
Groups:
- CR Flex Fixed Bearing Knee: Study arm will consist of patients that are treated with the NexGen CR-Flex Fixed Bearing Knee.
- CR Standard Knee: Study arm will consist of patients that are treated with the NexGen CR Knee.
Period: Overall Study
Arm/Group | CR Flex Fixed Bearing Knee | CR Standard Knee
Started | 87 | 102
Completed | 52 | 48
Not Completed | 35 | 54
Not completed — Lost to Follow-up | 6 | 11
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Death | 0 | 1
Not completed — Adverse Event | 26 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CR Flex Fixed Bearing Knee | CR Standard Knee | Total
Number analyzed (Participants) | 87 | 102 | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 48 | 85
  >=65 years | 50 | 54 | 104
Age Continuous [Mean (Standard Deviation); unit: years] | 66.8 (8.5) | 65.7 (8.5) | 66.2 (189)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 48 | 101
  Male | 34 | 54 | 88
Region of Enrollment [Number; unit: participants]
  United States | 87 | 102 | 189

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Range of Motion (ROM)
Description: The subject will have the operative joint's range of motion/movement assessed through a series of exercises and bends. The assessor will measure how far the joint bends/moves in each direction by degrees. The measurements are taken at each visit interval and recorded.
Time Frame: 24 Months
Population: There was one case in the CR Standard Knee cohort where the Range of Motion was not complete. Therefore, the total number analyzed is 47 and not 48.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | CR Flex Fixed Bearing Knee | CR Standard Knee
Number analyzed (Participants) | 52 | 47
degrees | 119.1 (16.5) | 120.7 (11.1)

2. Secondary Outcome: Return to Function (RtF) Via Knee Scoiety Score (Modified)
Description: Scores were calculated from responses on a modified Knee Society Score by the enrolled subjects for the stated visit intervals.
  Grading for the Knee Society Score is based on a scale from 0-100 and results are estabalished follows: 80-100 = Excellent; 70-79 = Good; 60-69 = Fair; and Below 60 = Poor.
Time Frame: 24 Months
Population: There was one case in the CR Flex Fixed cohort and 3 in the CR Standard Knee cohort where the Return to Function was not complete. Therefore, the total number analyzed is 51 instead of 52 and 45 instead of 48 respectfully.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR Flex Fixed Bearing Knee | CR Standard Knee
Number analyzed (Participants) | 51 | 45
units on a scale | 80.9 (18.8) | 85.1 (16.9)

ADVERSE EVENTS:
Arm/Group | CR Flex Fixed Bearing Knee | CR Standard Knee
Serious Adverse Events (participants affected / at risk) | 1/87 | 2/102
Other Adverse Events (participants affected / at risk) | 2/87 | 6/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CR Flex Fixed Bearing Knee (N=87) | CR Standard Knee (N=102)
Death (General disorders) | 0 (0) | 1 (1)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Articular Polyethylene Excessive Wear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CR Flex Fixed Bearing Knee (N=87) | CR Standard Knee (N=102)
Other Knee Related Complication (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Stiff Knee Resulting in Manipulation (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No